CLINICAL TRIAL: NCT00712829
Title: A Phase I Study Evaluating the Safety, Pharmacokinetics, Tissue Distribution, Metabolism of Small Molecule Inhibitors of Prostate Specific Membrane Antigen: Determination of I-123 Radiation Dosimetry for 123-I-MIP-1072 and 123-I-MIP-1095
Brief Title: Study to Evaluate the Safety, Pharmacokinetics, Tissue Distribution, Metabolism and Dosimetry of Two Prostate Cancer Imaging Agents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Molecular Insight Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: TX-P101
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Imaging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 123-I-MIP-1072 administration followed by 123-I-MIP-1095 administration two weeks later.
  Interventions: Drug: 123-I-MIP-1072; Drug: 123-I-MIP-1095
- 2 (Experimental): 123-I-MIP-1095 administration followed by 123-I-MIP-1072 administration two weeks later.
  Interventions: Drug: 123-I-MIP-1072; Drug: 123-I-MIP-1095

INTERVENTIONS:
Drug: 123-I-MIP-1072 — 10 mCi intravenous injection given one time during the study
Drug: 123-I-MIP-1095 — 10 mCi intravenous injection given one time during the study

SUMMARY:
This is a single blinded, randomized, cross-over design. Up to 12 patients will be randomly administered a single 10.0 mCi dose of 123I-MIP-1072 or 123I-MIP-1095 (study drugs). The second (alternate) study drug will be administered approximately 14 days after the first. A final follow-up visit will occur approximately 2 weeks after the injection of the alternate study drug.

ELIGIBILITY:
Inclusion Criteria:

* Have a prior histological diagnosis of prostate cancer.
* Have evidence of recurrent metastatic disease demonstrated by an abnormal bone scan, CT scan or MRI plus:

  1. PSA> 1.0 if patient is post prostatectomy or post ablative radiotherapy, or
  2. PSA> 20 if intact prostate
* Have platelet count of > 50,000/mm3
* Have neutrophil count of > 1,000/mm3
* Provide written informed consent and willing to comply with protocol requirements
* Greater than or equal to 18 years of age
* Can be on hormonal therapy if dose stable for > 90 days

Exclusion Criteria:

* Karnofsky performance status of <60
* Inadequate venous access (two antecubital or equivalent venous access sites are required for study drug injection and PK blood sampling, respectively)
* Patient received a permanent prostate brachytherapy implant within the last 3 months (for Pd-103 implants) or 12 months (for I-125 implants).
* Patient received external beam therapy or chemotherapy within the last 30 days
* Administered a radioisotope within 5 physical half lives prior to study enrollment
* Serum creatinine > 3.5 mg/dL
* Total bilirubin > 2.5 times the upper limit of normal
* Liver transaminases greater than 5x the upper limit of normal
* Received an investigational compound and/or medical device or is part of an investigational study within the past 30 days before enrollment into this study
* Have any medical condition or other circumstances which, in the opinion of the Investigator, would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study and/or post dose follow-up examinations
* Is determined by the Investigator that the patient is clinically unsuitable for the study
* Have had any other malignancies within 5 years other than basal or squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To examine the pharmacokinetics and organ radiation dosimetry of 123-I-MIP-1072 and 123I-MIP-1095 in patients with prior histological diagnosis of prostate cancer with evidence of recurrent metastatic disease.

SECONDARY OUTCOMES:
To examine whole body excretion and metabolism of 123-I-MIP-1072 and 123-I-MIP-1095 in patients with recurrent metastatic prostate cancer.
To evaluate the safety of administering a 10.0 mCi dose of 123-I-MIP-1072 and 123-I-MIP-1095 to patients with recurrent metastatic prostate cancer.
Optimize imaging parameters

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Johns Hopkins Medical Institutes - Neuroradiology Division, Baltimore, Maryland
  - New York Weill Cornell Medical Center - New York Presbyterian Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina